CLINICAL TRIAL: NCT05025072
Title: A Bioequivalence Study to Compare the Pharmacokinetics of Two Formulations of Siklos® in Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Theravia (Industry)
Collaborators: Simbec-Orion Group (Industry); Oncodesign SA (Industry); PhinC Development (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: SIK-FR-21-1
Record Dates: First submitted 2021-08-05; First posted 2021-08-27 (Actual); Last update posted 2021-10-07 (Actual); Status verified 2021-10

CONDITIONS: Healthy Volunteers
Keywords: Hydroxycarbamide; Hydroxyurea
MeSH Terms: interventions — Hydroxyurea

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Test IMP (Experimental): Hydroxycarbamide dispersible tablets (20 x 50 mg)
  Interventions: Drug: Hydroxycarbamide dispersible tablets; Drug: Hydroxycarbamide film-coated tablet
- Reference IMP (Active Comparator): Hydroxycarbamide film-coated tablet (1000 mg)
  Interventions: Drug: Hydroxycarbamide dispersible tablets; Drug: Hydroxycarbamide film-coated tablet

INTERVENTIONS:
Drug: Hydroxycarbamide dispersible tablets — Hydroxycarbamide dispersible tablets (20 x 50 mg)
Drug: Hydroxycarbamide film-coated tablet — Hydroxycarbamide film-coated tablet (1000 mg)

SUMMARY:
This study is a Phase I, open-label, single-centre, randomised, two-period, single-dose crossover study to compare and assess the bioequivalence, safety, tolerability and pharmacokinetics of hydroxycarbamide dispersible tablets (20 x 50 mg) (test IMP) and Siklos® film-coated tablet (1000 mg) (reference IMP) following single-dose administration. Thirty (30) healthy male and female participants, between 18 and 50 years of age are planned to participate in the study.

Study participants will be randomised to one of the 2 possible combination sequences. After each treatment administration, blood samples will be collected at specific time points to assess the Pharmacokinetics (PK) parameters.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy male and female participants, between 18 and 50 years of age, inclusive.
2. Female participant of childbearing potential willing to use a highly effective method of contraception, if applicable from the first dose until 3 months after the last dose of IMP.
3. Female participant of non-childbearing potential. For the purposes of this study, this is defined as the participant being amenorrhoeic for at least 12 consecutive months or at least 4 months post-surgical sterilisation.
4. Female participant with a negative pregnancy test at Screening.
5. Male participant (and partner of child bearing potential) willing to use a highly method of contraception, if applicable from first dose until 3 months after last dose of IMP.
6. Participant with a BMI of 18-29.9 kg/m2.
7. No clinically significant history of previous allergy / sensitivity to hydroxycarbamide or any of the excipients contained within the IMP(s).
8. No clinically significant abnormal test results for serum biochemistry, haematology and/or urine analyses within 28 days before the first dose administration of the IMP.
9. Participant with a negative urinary DOA screen (including alcohol) test results, determined within 28 days before the first dose administration of the IMP.
10. Participant with negative human immunodeficiency virus (HIV), hepatitis B surface antigen (HBsAg) and hepatitis C virus antibody (HCV Ab) test results at Screening.
11. No clinically significant abnormalities in 12-lead ECG determined within 28 days before the first dose of IMP.
12. No clinically significant abnormalities in vital signs determined within 28 days before the first dose of IMP.
13. Participant must be available to complete the study.
14. Participant must satisfy an Investigator about his/her fitness to participate in the study.
15. Participant must provide written informed consent to participate in the study.

Exclusion Criteria:

1. A clinically significant history of gastrointestinal disorder likely to influence IMP absorption.
2. Use of prescription or non-prescription drugs, including vitamins, herbal and dietary supplements within 28 days or 5 half-lives prior to the first dose of IMP.
3. Evidence of renal, hepatic, central nervous system, respiratory, cardiovascular, or metabolic dysfunction.
4. A clinically significant history of drug or alcohol abuse within the past two years.
5. Inability to communicate well with the Investigators.
6. Participation in a New Chemical Entity clinical study within the previous 3 months or five half-lives whichever is the longest, or a marketed drug clinical study within the 30 days or five half-lives whichever is the longest, before the first dose of IMP.
7. Donation of 450 mL or more blood within the 3 months before the first dose of IMP.
8. Users of nicotine products i.e., current smokers or ex-smokers who have smoked within 6 months prior to Screening or users of cigarette replacements
9. Female participants who are pregnant, breastfeeding or lactating.
10. Participants who have received any live or attenuated vaccine within 28 days of the first dose of IMP, or who are planning to receive a vaccine up to 28 days after receiving the last dose of IMP in Treatment Period 2.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 28 (Actual)
Dates: Start 2021-08-22 (Actual); Primary Completion 2021-09-29 (Actual); Study Completion 2021-09-29 (Actual)

PRIMARY OUTCOMES:
Cmax | 24 hours
  The observed maximum concentration (Cmax) in plasma
AUC0-t | 24 hours
  The area under the plasma concentration-time curve from time zero (pre-dose) to the time of last quantifiable concentration (t)
AUC0-infinity | 24 hours
  The AUC from time 0 to infinity

SECONDARY OUTCOMES:
tmax | 24 hours
  The time at which Cmax is apparent
t1/2 | 24 hours
  The terminal elimination half-life
ke | 24 hours
  The terminal elimination rate-constant
AUC%extra | 24 hours
  % of AUC0-infinity extrapolated
Adverse events | 24 hours
  Incidence of Adverse Events

CONTACTS AND LOCATIONS:
Overall Officials: Annelize Koch, MD, Principal Investigator — Simbec-Orion Group
Locations (1):
- Simbec-Orion Clinical Pharmacology, Merthyr Tydfil, United Kingdom

IPD SHARING:
Plan to Share IPD: No